CLINICAL TRIAL: NCT04890548
Title: A Mechanistic Study to Evaluate the Vasodilatory Effects of AZD3427 in Patients With Heart Failure With Preserved Ejection Fraction (HFpEF) and Patients With Heart Failure With Reduced Ejection Fraction (HFrEF)
Brief Title: Study to Evaluate the Effects of AZD3427 in Patients With Heart Failure
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Study start up timelines delayed into late autumn, and with COVID cases rising in the UK, the feasibility of successfully recruiting the study and ethical concerns about starting a study that AZ may not be able to complete.
Sponsor: AstraZeneca (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D8330C00002
Record Dates: First submitted 2021-05-13; First posted 2021-05-18 (Actual); Last update posted 2021-12-17 (Actual); Status verified 2021-12

CONDITIONS: Heart Failure
Keywords: Heart Failure with Preserved Ejection Fraction; Heart Failure with Reduced Ejection Fraction; Forearm blood flow
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with HFpEF or HFrEF (Experimental): Patients will be enrolled in 2 cohorts in parallel: 1 cohort of patients with HFpEF and 1 cohort of patients with HFrEF. Patients will receive a sequence of 5 IA infusions into the brachial artery, consisting of a baseline saline infusion of approximately 20 minutes, followed by 3 sequential infusions of AZD3427 at ascending doses of approximately 10 minutes (each) and a washout saline infusion of approximately 15 minutes.
  Interventions: Drug: AZD3427

INTERVENTIONS:
Drug: AZD3427 — Patients will receive 5 IA infusions of AZD3427 into the brachial artery. The IA infusions of AZD3427 will be administered via a syringe pump, using a polypropylene syringe containing 0.9% (w/v) saline and delivered through an administration set comprising a syringe, extension tubing (PVC), and a 0.2- or 0.22-μm PVDF syringe filter.

SUMMARY:
The primary purpose of this mechanistic study is to evaluate the vasodilatory effects of AZD3427 in adult patients with heart failure and will be performed at approximately 2 study sites in the United Kingdom.

DETAILED DESCRIPTION:
The study will enroll patients in 2 cohorts in parallel: 1 cohort of patients with heart failure with preserved ejection fraction (HFpEF) and 1 cohort of patients with heart failure with reduced ejection fraction (HFrEF). Each cohort plans to enroll at least 7 evaluable patients.

All patients will receive the same sequence of 5 intra-arterial (IA) infusions into the brachial artery, consisting of a baseline saline infusion of approximately 20 minutes, followed by 3 sequential infusions of AZD3427 at ascending doses of approximately 10 minutes (each) and a washout saline infusion of approximately 15 minutes.

For each patient, the study will last at least 51 days and up to 99 days, including:

* A screening period of 1 to 42 days (which will include baseline echocardiography)
* A single-day treatment period during which patients will stay at study site until at least 4 hours after the end of infusions
* A follow-up period of 49 to 56 days after the end of the last infusion including:

A follow-up phone call on Day 2 (within 24 ± 6 hours post-infusion) A follow-up visit on Day 8 (+ 3 days) A follow-up visit on Day 29 (± 2 days) A follow-up visit on Day 50 (+ 7 days)

ELIGIBILITY:
Inclusion Criteria:

1. Patient must be 18 to 75 years of age.
2. Patient with known clinical diagnosis of Stage C heart failure New York Heart Association (NYHA) Class I-III and on stable medical therapy for at least 12 weeks prior to screening with no significant dose change or new medications added during that period. Specifically:

   1. Patients with a diagnosis of HFrEF, defined as ejection fraction ≤ 40%. OR
   2. Patients with a diagnosis of HFpEF, defined as ejection fraction ≥ 50%.
3. Patients with suitable veins and arteries for cannulation or repeated puncture.
4. Patients who are able to lie flat for the duration of IA infusions and related procedures during Visit 2 (approximately 3 hours).
5. Body weight of at least 60 kg and body mass index within the range of 18 to 40 kg/m^2.
6. Male and/or female of nonchildbearing potential.
7. Capable of giving signed informed consent.

Exclusion Criteria:

1. History of any clinically important disease or disorder which, in the opinion of the investigator, may either put the participant at risk because of participation in the study, or influence the results or the participant's ability to participate in the study.
2. Clinically significant valvular heart disease as judged by the investigator.
3. Congenital heart disease (patients with Patent Foramen Ovale may be included in the study).
4. Clinical diagnosis of heart failure NYHA Class IV.
5. Occurrence in the last 3 months of any of the following:

   1. Acute coronary syndrome: myocardial infarction or unstable angina.
   2. Percutaneous coronary intervention.
   3. Cerebrovascular accident or transient ischaemic attack.
   4. Heart failure hospitalisation.
6. History of prior dissections.
7. History or suspicion of cardiac amyloidosis.
8. Patients with conditions where vasodilator therapy may be contraindicated.
9. History of cancer in the last 5 years, except for non-melanoma skin cancer.
10. Any clinically important abnormalities in clinical chemistry, haematology or urinalysis.
11. Any positive result at Screening for serum hepatitis B surface antigen, hepatitis C antibody and human immunodeficiency virus.
12. History of severe allergy/hypersensitivity or ongoing clinically important allergy/hypersensitivity, as judged by the investigator.
13. Abnormal vital signs, after at least 10-minute supine rest, defined as any of the following at Screening:

    1. Systolic blood pressure (BP) > 160 mmHg.
    2. Diastolic BP > 90 mmHg.
14. Any clinically important abnormalities in rhythm, conduction or morphology of the resting 12-lead electrocardiogram as considered by the investigator.

    1. Prolonged QTcF > 450 ms.
    2. Family history of long QT syndrome.
    3. Second or third-degree AV block, or sinus node dysfunction with significant sinus pause.
15. History of hypersensitivity to drugs with a similar chemical structure or class to AZD3427.
16. Participants who have previously received AZD3427.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-11-23 (Estimated); Primary Completion 2022-08-02 (Estimated); Study Completion 2022-08-02 (Estimated)

PRIMARY OUTCOMES:
Maximum change from baseline in absolute forearm blood flow in the infused arm during AZD3427 IA infusions | Day 1
  To determine whether AZD3427 produces a vasodilatory response in the forearm resistance vessels of HFpEF and HFrEF patients, as assessed by forearm blood flow parameters measured using venous occlusion plethysmography.

SECONDARY OUTCOMES:
Number of patients with anti-drug antibody (ADAs) in serum samples at baseline and at Day 8, Day 29, and Day 50 | Day 1, Day 8, Day 29 and Day 50
  To assess the immunogenicity of AZD3427.
Change from baseline in forearm blood flow ratio in the infused arm (AZD3427 infusion:baseline) after each AZD3427 IA infusion | Day 1
  To determine whether AZD3427 produces a vasodilatory response in the forearm resistance vessels of HFpEF and HFrEF patients, as assessed by forearm blood flow parameters measured using venous occlusion plethysmography.
Change from baseline in forearm blood flow ratio between arms (infused arm:non-infused arm) after each AZD3427 IA infusion | Day 1
  To determine whether AZD3427 produces a vasodilatory response in the forearm resistance vessels of HFpEF and HFrEF patients, as assessed by forearm blood flow parameters measured using venous occlusion plethysmography.

OTHER OUTCOMES:
Number of patients with adverse events | From Screening (Day -42 to Day -1) until the Follow-up visit (Day 1, Day 2, Day 8, Day 29, and Day 50)
  Assessment of safety and tolerability of AZD3427 in HFpEF and HFrEF patients, following low-dose local IA infusion of 3 sequential ascending doses of AZD3427.

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All requests will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please refer to our disclosure commitment at: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool. Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home